CLINICAL TRIAL: NCT04966130
Title: Effect of Urinary Indwelling Time on Early Continence After Robot-assisted Radical Cystectomy With Orthotopic Ileal Neobladder.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SysMU-RARC1
Record Dates: First submitted 2021-07-09; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Muscle-Invasive Bladder Carcinoma
Keywords: muscle-invasive bladder cancer; robot-assisted radical cystectomy; urinary indwelling time; continence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The clinical trial assesses the effect of urinary indwelling time on early continence after robot- assisted radical cystectomy with orthotopic ileal neobladder.

DETAILED DESCRIPTION:
Radical cystectomy is the gold standard for muscle-invasive bladder. Orthotopic ileal neobladder, as one of the urinary diversion methods, is preferred whenever possible to achieve a better postoperative quality of life. After surgery, the patient usually indwells a catheter until the anastomotic site heals. And the urinary indwelling time may have an effect on early continence. This is a prospective study including patients undergoing RARC with orthotopic ileal neobladder. Urinary continence recovery and perioperative complication will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed bladder cancer
2. Undergoing robot-assisted radical cystectomy with orthotopic ileal neobladder
3. Complete perioperative clinical data

Exclusion Criteria:

1. Patients diagnosed with distant metastasis
2. Patients who had urinary incontinence before surgery
3. Patients with unavailable follow-up data

Ages: 18 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients undergoing robot- assisted radical cystectomy with orthotopic ileal neobladder will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Day-time continence rate | 1 year
Night-time continence rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University